CLINICAL TRIAL: NCT03424317
Title: Evaluation of the Therapeutic Effect of Sodium Intake Reduction by Education in Patients With Treatment Resistant Hypertension
Brief Title: Therapeutic Effect of Sodium Intake Reduction in Treatment Resistant Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult in recruitment, frequent withdrawal
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Moo-Yong Rhee, Proffessor, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUMC-C1701
Record Dates: First submitted 2017-11-16; First posted 2018-02-07 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Sodium Intake; Resistant Hypertension
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: single blind, randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium intake reduction and exercise (Active Comparator): education of sodium intake reduction and regular exercise
  Interventions: Behavioral: Sodium intake reduction; Behavioral: Exercise
- Exercise (Placebo Comparator): education of regular exercise only
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Sodium intake reduction — Provide materials to reduce sodium intake and educate how to reduce sodium intake effectively
  Arms: Sodium intake reduction and exercise
Behavioral: Exercise — Provides materials on exercise methods to reduce blood pressure and educates how to perform exercise effectively

SUMMARY:
The aim of this study was to evaluate the therapeutic effect of sodium intake reduction by education in patients with resistant hypertension.

The study was designed to maximize the compliance to antihypertensive agents and use optimal doses of antihypertensive agents including diuretics for 2 months before randomization. Patients will be assigned randomly to receiving (1) education of sodium intake reduction and exercise, or (2) education of exercise alone. Education of sodium intake reduction will be blinded to patients, and education of exercise will be provided to both group to blind the subjects. Daytime ambulatory blood pressure is adopted for diagnosis of resistant hypertension to avoid white-coat effect.

DETAILED DESCRIPTION:
The study consists of 3 phases. The first phase is to exclude pseudo-resistant hypertension by improving compliance to antihypertensive medications. Patients should visit with a prescribed antihypertensive drugs to calculate compliance to medication. If patient has compliance to medication >= 85% [= (the number of pills dispensed - the number of pills counted) / the number of pills expected to have been taken (calculated by multiplying the daily dose by the number of days since the date dispensed)], ambulatory blood pressure will be measured.

If the patient had compliance to medication >= 85%, and daytime ambulatory blood pressure >=135/85 mmHg, he will be entered into first phase of treatment. If patient had compliance to medication <85%, patients will be asked to enhance medication adherence to 85% or more, and revisit after 1 months.

In the first phase of treatment, dose of current antihypertensive medications (diuretics should be included) will be escalated to optimal doses. Three or more classes of antihypertensive drugs should be prescribed, and educate to keep compliance to medication >=85%. The duration of second phase of treatment is 2 months. After start of first phase, there is a monitoring visit monitoring of adverse drug reaction of diuretics for safety. If there is adverse drug reaction, the dose of suspected drug will be decreased. After 2 months of treatment, if daytime ambulatory blood pressure is >= 135/85 mmHg with compliance to medication >=85%, the patients will be entered into second phase of treatment.

In the second phase of treatment, patients will be randomly assigned to receive either education of exercise or education of exercise and low sodium diet (intensive education with education materials). To the patients assigned to exercise education, detailed training of diet control using educational materials will not be provided. The patients will be blinded to educational group assignments. The duration of second phase of treatment is 1 month. Before start and after completion of second phase of treatment, the amount of sodium intake will be measured by 24-hour urine sodium excretion.

ELIGIBILITY:
Inclusion Criteria:

* individuals who agreed to participate in the study and submitted written informed consent
* individuals aged 20 or more years
* Hypertensive patients whose blood pressure is not controlled normally while taking three or more antihypertensive agents including diuretics
* Diuretics should be Hydrochlorothiazide or Indapamide

Exclusion Criteria:

* Systolic blood pressure ≥ 220 mmHg
* Chronic kidney disease: estimated Glomerular filtration rate by Modification of Diet in Renal Disease formula ≤ 30 mL/min
* Hyperkalemia (>5.5 mmol/L) or hypokalemia (<3.5 mmol/L)
* Hyponatremia (<135 mmol/L)
* Major cardiovascular events (MI, unstable angina, coronary revascularization, stroke) within 6 month of screening
* Retinal bleeding within 3 months
* Heart failure stage 3 or 4
* Severe liver disease
* Pregnancy or women in the fertile age not using efficient contraceptive methods
* Alcoholism
* Renovascular disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Difference of change of sitting systolic blood pressure | from randomization to completion of second phase of treatment (sodium intake reduction phase, for 1 month)
  Comparison of the difference of sitting systolic blood pressure after completion of second phase of treatment (sodium intake reduction phase) from randomization of Second phase of treatment between groups

SECONDARY OUTCOMES:
Effect of optimized antihypertensive treatment | At the end of First phase of treatment (for 2 months)
  Percent of responders (sitting SBP < 90 mmHg or difference of sitting SBP > 10 mmHg from randomization) at the end of first phase treatment
Effect of optimized antihypertensive treatment | From the start to the end of First phase of treatment (for 2 months)
  Comparison of changes of systolic and diastolic blood pressure lowering at the end of the First phase of treatment from baseline
Effect of sodium intake reduction | from randomization to completion of second phase of treatment (sodium intake reduction phase, for 1 month)
  Difference of change of sitting diastolic blood pressure between groups (exercise vs exercise + sodium intake reduction) after completion of the Second phase of treatment (sodium intake reduction phase) from randomization of Second phase of treatment
Comparison of Percent of responders at the end of first phase treatment between groups | at the end of second phase of treatment (sodium intake reduction phase, for 1 month)
  Comparison of percent responders between groups (sitting SBP < 90 mmHg or difference of sitting SBP > 10 mmHg from randomization) at the end of second phase of treatment

OTHER OUTCOMES:
Difference of renin and aldosterone level between non-resistant hypertension vs resistant hypertension | after completion of first phase treatment (2 months)
  Comparison of renin and aldosterone level between non-resistant hypertension vs resistant hypertension after optimized antihypertensive treatment
Difference of the effect of sodium intake reduction on renin and aldosterone level between responders vs non-responders to sodium intake reduction | after completion of second phase treatment (1 month)
  Comparison of renin and aldosterone level between responders vs non-responders to sodium intake reduction
Effect of compliance improvement in BP control | Phase of improving drug adherence (1 month)
  Effect of compliance improvement in BP control

CONTACTS AND LOCATIONS:
Overall Officials: Moo-Yong Rhee, MD, Principal Investigator — Dongguk University Ilsan Hospital/Cardiovascular Center
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
The study data will be shared with investigators who will participate this study as primary investigator or sub-investigator.